CLINICAL TRIAL: NCT00911222
Title: Epidemiologic Registry for the Description of Antiemetic Strategies Under Real-life Conditions.
Brief Title: Epidemiological EMESIS-Registry
Acronym: EMESIS
Status: Completed | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Collaborators: Arbeitsgemeinschaft fur Internistische Onkologie (Other); ASORS (Unknown); Arbeitskreis Klinische Studien (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: IOM-143; IOM-143
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Antiemetic Therapy
Keywords: antiemetic therapy; emesis; vomiting; nausea; moderately and highly emetogenic chemotherapy; cisplatin; carboplatin; oxaliplatin; anthracycline; cyclophosphamid
MeSH Terms: conditions — Vomiting; Nausea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- antiemetic treatment: epidemiological registry
  Interventions: Other: non-interventional

INTERVENTIONS:
Other: non-interventional — non-interventional

SUMMARY:
The purpose of this registry is to record information on reality of anti-emetic therapies of cancer-patients in Germany. The outcome of this study is the efficacy of anti-emetic therapies dependent on the rate "complete and major control" of nausea and emesis in moderately and highly emetogenic chemotherapies, consisting of platin-derivates (cisplatin, carboplatin and oxaliplatin), anthracyclines and/or cyclophosphamid.

ELIGIBILITY:
Inclusion Criteria:

* Moderately or highly emetogenic chemotherapy consisting of platin-derivates (cisplatin, carboplatin and oxaliplatin), anthracyclines and/or cyclophosphamid.
* start with the 1st cycle of the regimen (chemo naive patients). Inclusion of pretreated patients is also possible, if the last treatment cycle of a previous chemotherapy was given >= 24 months ago.
* Compliance with registry procedures
* Age >= 18 years
* WHO Performance Status of 0 or 1 (Karnofsky-Index >= 70%)
* Life expectancy of at least 12 weeks
* Signed and dated informed consent before the start of the registry

Exclusion Criteria:

* Mentally incapable or incompliant patients
* Last chemotherapy <= 24 months (if pretreated)
* Known hypersensitivity to antiemetic medication
* unability of the patient to be treated with oral medication
* pregnancy or lactation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Practitioners specialized in oncology, hematology and/or gynaecology
Sampling Method: Non-Probability Sample
Enrollment: 1035 (Actual)
Dates: Start 2008-10; Primary Completion 2009-05 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Efficacy of anti-emetic therapies dependent on the rate "complete and major control" of nausea and emesis in moderately and highly emetogenic chemotherapy regimens. | 4 chemotherapy applications per patient

CONTACTS AND LOCATIONS:
Overall Officials: Jan Schröder, Dr. med. / MD, Principal Investigator — Praxis für Hämatologie und Onkologie
Locations (1):
- iOMEDICO AG, Freiburg im Breisgau, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] American Society of Clinical Oncology; Kris MG, Hesketh PJ, Somerfield MR, Feyer P, Clark-Snow R, Koeller JM, Morrow GR, Chinnery LW, Chesney MJ, Gralla RJ, Grunberg SM. American Society of Clinical Oncology guideline for antiemetics in oncology: update 2006. J Clin Oncol. 2006 Jun 20;24(18):2932-47. doi: 10.1200/JCO.2006.06.9591. Epub 2006 May 22. PMID 16717289
- [Background] MASCC guidelines: Consensus Conference on Antiemetic Therapy, Perugia, march 29 - 31. 2004, update: December 2007)
- [Background] Osoba D, Zee B, Warr D, Kaizer L, Latreille J, Pater J. Quality of life studies in chemotherapy-induced emesis. Oncology. 1996 Jun;53 Suppl 1:92-5. doi: 10.1159/000227647. PMID 8692559
- [Background] Laszlo J, Lucas VS Jr. Emesis as a critical problem in chemotherapy. N Engl J Med. 1981 Oct 15;305(16):948-9. doi: 10.1056/NEJM198110153051609. No abstract available. PMID 7278899
- [Background] Gralla RJ. Controlling emesis in patients receiving cancer chemotherapy. Recent Results Cancer Res. 1991;121:68-85. doi: 10.1007/978-3-642-84138-5_9. No abstract available. PMID 1857886
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716